CLINICAL TRIAL: NCT01539590
Title: A Phase 2 Pilot Study to Evaluate the Safety and Activity of BB3 as an Adjunct to Percutaneous Coronary Intervention (PCI) in Subjects Presenting With Acute ST Segment Elevation Myocardial Infarction (STEMI)
Brief Title: Study to Evaluate the Safety and Activity of BB3 to Treat Heart Attack
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001-10; 5R44HL091699 (NIH)
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Myocardial Infarction
Keywords: hepatocyte growth factor mimetic; hepatocyte growth factor(HGF); Myocardial Infarction; Acute ST Segment Elevation Myocardial Infarction (STEMI); Percutaneous Coronary Intervention (PCI)
MeSH Terms: conditions — Myocardial Infarction; Deafness, Autosomal Recessive 39; ST Elevation Myocardial Infarction | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BB3 (Experimental): Daily intravenous administration of 2 mg/kg BB3 for four (4) days
  Interventions: Drug: BB3
- Normal Saline (Placebo Comparator): Daily intravenous administration for four (4) days
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: BB3 — Daily intravenous administration of 2 mg/kg BB3 for four (4) days
  Arms: BB3
Drug: Normal saline — Daily intravenous administration for four (4) days. The volume of normal saline will vary by estimated weight.
  Arms: Normal Saline

SUMMARY:
The study will evaluate the effect of BB3 to preserve myocardial (heart) tissue and function following myocardial infarction (heart attack).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) has become the mainstay for treatment of ST-segment elevation myocardial infarction (STEMI). Whereas early recanalization undoubtedly salvages myocardial tissue, reperfusion following prolonged ischemia can also exacerbate injury. Infarct size needs to be limited, and the conditions favoring adaptive ventricular healing and remodeling optimized because in patients with acute myocardial infarction (AMI) who do not die of out-of-hospital arrhythmias, long-term prognosis is dependent on the amount of myocardium that is lost, and the outcome of ventricular remodeling. Angion Biomedical Corp. has identified BB3, a small molecule mimetic of hepatocyte growth factor/scatter factor (HGF/SF) whose activity is expected to preserve tissue viability and attenuate dysfunction in the setting of organ injury while obviating the logistical difficulties associated with gene or protein therapy. HGF/SF is a naturally occurring cell survival factor that holds significant therapeutic potential. BB3 has been shown to possess HGF/SF activities, including protection against heart injury following myocardial infarction. This study is designed to evaluate clinical efficacy of BB3 in patients presenting with acute ST segment elevation myocardial infarction (A-STEMI) who undergo PCI.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has been provided and signed written informed consent, approved by the Institutional Review Board (IRB), prior to performance of any study related procedure including screening procedure.
2. Subject is male or female
3. Subject is 21 to 80 years of age
4. Estimated body weight < 120 kg and BMI < 40
5. Subject is experiencing clinical symptoms consistent with acute myocardial infarction (AMI) (e.g., chest pain, arm pain, etc.,) >30 minutes duration and unresponsive to nitroglycerin; with ST segment elevation of more than 1 mm in at least two contiguous leads of ECG or new or presumed new onset bundle branch block (BBB)
6. Fulfills clinical center's criteria for primary PCI
7. PCI will be done within 12 hours of onset of STEMI.
8. The subject and his/her physician are willing to comply with the requirements of the study and the specified follow-up evaluations.
9. If female, either surgically sterile or post-menopausal or using acceptable contraception and agree to use effective birth control regimen during the study period. Men must agree to use condoms during the study period. Women of child bearing potential must have a negative urine or serum pregnancy test.
10. In the opinion of the Investigator, the subject is capable of understanding and complying with the protocol.

Exclusion Criteria:

1. Pregnant or nursing subjects and those who plan pregnancy in the period up to 6 months following index procedure.
2. Cardiogenic shock (Killip class 4) or cardiac arrest
3. History of prior myocardial infarction or pre-existing Q waves on ECG
4. An elective surgical procedure is planned that would necessitate interruption of anti-platelet agents during the first six months post enrollment;
5. Any contraindication to undergo MRI imaging. This will include any of the following exclusions:

   1. Cardiac pacemaker or implantable defibrillator;
   2. Non-MRI-compatible aneurysm clip;
   3. Neural stimulator (e.g., TENS-Unit);
   4. Any implanted or magnetically activated device (e.g., insulin pump);
   5. Any type of non-MRI-compatible metallic ear implant;
   6. Metal shavings in the orbits;
   7. Any metallic foreign body, shrapnel, or bullet in a location which the physician feels would present a risk to the subject;
   8. Any history indicating contraindication to MRI, including claustrophobia or allergy to gadolinium;
   9. Inability to follow breathhold instructions or to maintain a breathhold for >15 seconds;
   10. Irregular cardiac rhythm not expected to resolve after treatment of the acute cardiac condition (e.g., chronic atrial fibrillation)
   11. Known hypersensitivity or contraindication to gadolinium contrast.
6. Subject has active bleeding or a history of bleeding diathesis or coagulopathy (including heparin induced thrombocytopenia), or refusal to receive blood transfusions if necessary;
7. Subjects presenting with cardiogenic shock (SBP <80 mmHg for >30 minutes, or requiring IV pressors or emergency IABP for hypotension treatment) or cardiopulmonary resuscitation prior to randomization;
8. History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke; stroke or transient ischemic attack within the past 6 months, or any permanent residual neurologic defect; known preceding cardiac ventricular arrhythmia
9. Impaired renal function (eGFR of ≤30 ml/min/1.73m2, as estimated by the MDRD4v equation) or on dialysis.
10. Impaired hepatic function (ALT > 2x upper limit of normal, or a total bilirubin greater than 1.5 x upper limit of normal).
11. Currently participating in or has participated in an investigational drug or medical device study within 30 days or 5 half-lives, whichever is longer, prior to enrollment into this study
12. Have an active malignancy or history of solid, metastatic, or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed
13. History of positive human immunodeficiency virus (HIV) test
14. History of rheumatoid arthritis
15. History of proliferative retinopathy or laser surgery for retinopathy
16. Subjects who require cytochrome P450 1A2 (CYP1A2) inhibitors, ciprofloxacin and/or fluvoxamine (Luvox®)
17. Subject has other medical illness or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy of less than 6 months,
18. Any significant medical condition which in the Investigator's opinion may interfere with the subject's optimal participation in the study;
19. Subject has a known hypersensitivity or allergy to stainless steel, nickel, cobalt chromium, nitinol, titanium or known hypersensitivity or allergy to contrast media (e.g. rash) that cannot effectively be controlled by premedication with steroids and/or diphenhydramine. Subjects with hypersensitivity or allergy to any of the components of the device (structural, drug or polymer components) and subjects with true prior anaphylaxis to contrast media should not be enrolled

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weizhong Cai, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Yale University Medical Center, New Haven, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- BB3, 4 Daily Doses: BB3: Daily intravenous administration of 2 mg/kg BB3 for four (4) days ; 10 to 12 minutes; small molecule mimetic of hepatocyte growth factor
- Placebo; 4 Daily Doses: Placebo: Normal saline; Daily intravenous administration for four (4) days. The volume of normal saline will vary by estimated weight.
Period: Overall Study
Arm/Group | BB3, 4 Daily Doses | Placebo; 4 Daily Doses
Started | 3 | 2
Complete Study Treatment | 1 | 2
Completed | 0 | 2
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- BB3, 4 Daily Doses: BB3: Daily intravenous administration of 2 mg/kg BB3 for four (4) days
- Placebo: Normal saline. Daily intravenous administration for four (4) days.
- Total: Total of all reporting groups
Arm/Group | BB3, 4 Daily Doses | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 61 [50 to 75] | 57.5 [46 to 69] | 59 [46 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Reduction in Infarct Size
Description: Evaluation of reduction in infarct size by MRI between the BB3 and placebo treatment groups at 6 months based on index of myocardial salvage
Time Frame: 6 month
Population: Five subjects were enrolled into the study; 3 subjects were randomized to BB3 and 2 subjects to placebo. Of the 3 subjects randomized to BB3, 1 completed study treatment; all three subjects discontinued the study prematurely. The two subjects randomized to placebo completed study treatment and neither discontinued the study prematurely.
Groups:
- Placebo, 4 Daily Doses: Normal saline. Daily intravenous administration for four (4) days.
Arm/Group | BB3, 4 Daily Doses | Placebo, 4 Daily Doses
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Evaluation of the Degree of Late Ventricular Remodeling
Description: Evaluation of the degree of late ventricular remodeling between the BB3 and placebo treatment groups at 6 months, as measured by increase in LV end-diastolic volume index (LVEDVI) from initial MR image (day 5±1) to late MR image (6 months).
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in CK-MB and Troponin
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in BNP Levels
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Symptoms and Clinical Signs of CHF
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in LVEDVI, LVESVI and LV Ejection Fraction (EF) After MI Assessed by Cine MR (SSFP Imaging)
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: LVEDVI, LVESVI and LVEF After MI Assessed by 2D and 3D Echocardiography
Time Frame: 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Change Between Initial Semi-quantitative Regional Wall Motion Score (17 Segment Model) by Echocardiography
Time Frame: 1 and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Regional Myocardial Radial, Circumferential and Longitudinal Strain
Time Frame: 1 and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Frequency of MACE
Time Frame: 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Frequency of New Onset CHF Through 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Number of Hospitalizations for CHF Through 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

13. Secondary Outcome: Incidence of Complete ST Segment Resolution 60 ± 30 Minutes After Last Angiogram
Time Frame: 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Frequency of AE, SAEs
Time Frame: 6 months
Reporting Status: Not Posted

15. Secondary Outcome: Frequency of MACCE
Time Frame: 6 months
Reporting Status: Not Posted

16. Secondary Outcome: All-cause Mortality
Time Frame: 6 months
Reporting Status: Not Posted

17. Secondary Outcome: Development of Ventricular Fibrillation or Other Life-threatening Arrhythmia
Time Frame: 6 months
Reporting Status: Not Posted

18. Secondary Outcome: Change From Baseline eCrCl
Time Frame: 6 months
Reporting Status: Not Posted

19. Secondary Outcome: Change in Body Weight
Time Frame: 6 months
Reporting Status: Not Posted

20. Secondary Outcome: Symptoms and Clinical Signs of CHF
Description: Symptoms and clinical signs of CHF measured by NYHA classification
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- BB3 Small Molecule Mimetic of Hepatocyte Growth Factor: small molecule mimetic of hepatocyte growth factor/scatter factor
  BB3: Daily intravenous administration of 2 mg/kg BB3 for four (4) days
- Placebo: Normal saline
  Placebo: Daily intravenous administration for four (4) days. The volume of normal saline will vary by estimated weight.
Arm/Group | BB3 Small Molecule Mimetic of Hepatocyte Growth Factor | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BB3 Small Molecule Mimetic of Hepatocyte Growth Factor (N=3) | Placebo (N=2)
bradycardia (Cardiac disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
headache (General disorders) | 0 | 1
hyperhidrosis (General disorders) | 1 | 0
nausea and vomiting (Gastrointestinal disorders) | 1 | 0
ventricular tachycardia (Cardiac disorders) | 1 | 0
dizziness (General disorders) | 1 | 0
infusion site pain (Surgical and medical procedures) | 1 | 0
tinnitus (Ear and labyrinth disorders) | 0 | 1
sinusitis (Infections and infestations) | 0 | 1
fatigue (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Five subjects were enrolled into the study; 3 subjects were randomized to BB3 and 2 subjects to placebo. All the 3 subjects randomized to BB3 discontinued the study prematurely. The 2 subjects randomized to placebo completed study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days